NCT NUMBER: DATE::10.08.25

## CONSENT OF THE RESPONDENT TO PARTICIPATE IN THE RESEARCH PROJECT

| Name of the re | search unit: |
|---|---|
| Name of the su | kiaat. |
| Name of the subject: | |
| Age | Address: |
| Name of the physician in charge of the research project: Contact phones for the respondent: | |
| Study topic: Evaluation of the efficacy of subgingival application of 1.2% lowastatin gel as an adjunct to conventional non-surgical therapy for periodontitis in generally healthy non-smoking and smoking patients from central Europe: a randomized split-mouth controlled trial. | |
| Name and last name of the subject: | |

## I hereby declare that:

- 1. I have been informed by the dentist about the purpose of the intended research and how it shall be conducted, and that I had the opportunity to ask questions of the research project leader and received answers to those questions.
- 2. I understand what the research project in which I have been invited to participate is about, and I understand that it is in the nature of a medical experiment.
- 3. I have familiarized myself with the contents of "Information for the patient participating in the study", of which I have received 1 copy.
- 4. I understand that I can refuse or revoke my consent to participate in the study at any time including during the course of the study, which will in no way affect my further treatment.

- 5. In the information to the respondent, I have been acquainted with the terms and conditions of insurance covering possible negative consequences of participation in the research project, and I accept these conditions. I received for review the policy from which they arise.
- 6. In consideration of the above I give my informed voluntary consent to participate in the research project and to process my data to the extent necessary for its implementation, however, subject to confidentiality preventing identification of my person by legal and natural persons other than those listed in the protocol as conducting the project and in accordance with *Information for the patient participating in the study*.
- 7. I received 1 copy of this document.

| Physician in charge of the research project: | Date: | Caption: |
|---|---|---|
| The respondent or his/her legal guardian: (insert appropriate) | Date: | Caption: |